CLINICAL TRIAL: NCT05300516
Title: Vagus Nerve-guided Versus Conventional Robotic-assisted Splenectomy and Azygoportal Disconnection
Brief Title: Vagus Nerve-guided Robotic-assisted Splenectomy and Azygoportal Disconnection
Acronym: VNRSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Clinical Professor, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YZUC-008
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Cirrhosis; Hypertension; Splenectomy; Robotic-assisted
Keywords: Vagus nerve; Delayed gastric emptying; Cirrhosis; Hypertension; Robotic-assisted
MeSH Terms: conditions — Fibrosis; Hypertension; Gastroparesis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vagus nerve-guided group (Experimental): Procedure/Surgery: vagus nerve-guided group The vagus nerve-guided procedure was performed in the following order: (1) find the left crural diaphragm; (2) via the surface of the left crural diaphragm, blunt dissect the left lateral surface of the distal esophagus using Bipolar Forceps, and find posterior vagal trunk; (3) along posterior vagal trunk towards left lateral esoph-agogastric junction, find and protect gastric and celiac branches; (4) enter the lesser omental sac from the right crural diaphragm using Bipolar Forceps; (5) transect the left gastric artery and vein together using a linear vascular stapler; (6) blunt dissect the anterior surface of the distal esophagus using Bipolar Forceps, and find anterior vagal trunk; (7) along anterior vagal trunk towards right lateral esoph-agogastric junction, find and protect gastric and hepatic branches; and (8) blunt dissect the right lateral surface of the distal esophagus. The hepatogastric ligament was conserved.
  Interventions: Procedure: vagus nerve-guided group
- Conventional group (No Intervention): Every patient of conventional group will receive the conventional Robotic-assisted azygoportal disconnection procedure.

INTERVENTIONS:
Procedure: vagus nerve-guided group — The vagus nerve-guided procedure was performed in the following order: (1) find the left crural diaphragm; (2) via the surface of the left crural diaphragm, blunt dissect the left lateral surface of the distal esophagus using Bipolar Forceps, and find posterior vagal trunk; (3) along posterior vagal trunk towards left lateral esoph-agogastric junction, find and protect gastric and celiac branches; (4) enter the lesser omental sac from the right crural diaphragm using Bipolar Forceps; (5) transect the left gastric artery and vein together using a linear vascular stapler; (6) blunt dissect the anterior surface of the distal esophagus using Bipolar Forceps, and find anterior vagal trunk; (7) along anterior vagal trunk towards right lateral esoph-agogastric junction, find and protect gastric and hepatic branches; and (8) blunt dissect the right lateral surface of the distal esophagus. The hepatogastric ligament was conserved.
  Arms: vagus nerve-guided group

SUMMARY:
This study aimed to evaluate whether vagus nerve-guided robotic-assisted splenectomy and azygoportal disconnection is effective and safe, and to determine whether a reduction in the incidence of postoperative complications of the digestive system improves postoperative quality of life compared with conventional robotic-assisted splenectomy and azygoportal disconnection.

DETAILED DESCRIPTION:
After successful screening the cases of cirrhosis of liver irrespective of the etiology who have non tumor portal vein thrombosis will be enrolled. The baseline parameter will be recorded and the patient will be randomized into either interventional (vagus nerve-guided robotic-assisted splenectomy and azygoportal disconnection) or control (conventional robotic-assisted splenectomy and azygoportal disconnection) group. From postoperative day 3, all patients will receive 2.5 mg oral Apixaban tablets (Bristol-Myers Squibb, Cruiserath, USA) twice daily for 6 months, low-molecular-weight heparin (CS Bio, Hebei, China) subcutaneously (4.100 IU/day) for 5 days, and 25 mg of oral dipyridamole (Henan Furen, Henan, China) thrice daily for 3 months. At months 3 after operation, electron gastroscopy examination for delayed gastric emptying will be done for all patients. Postoperative complications of the digestive system (including diarrhea, epigastric fullness, bloating, nausea, and vomiting), liver and renal function, and body weight will be recorded at the seventh day and months 3 after operation. Then 3 months monitoring will be done in the both groups as per the primary or secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical, radiological or histologic diagnosis of cirrhosis of any etiology
2. Splenomegaly with secondary hypersplenism
3. Bleeding portal hypertension
4. No evidence of portal vein system thrombosis by ultrasound evaluation and angio-CT
5. Informed consent to participate in the study

Exclusion Criteria:

1. Delayed gastric emptying
2. Diarrhea
3. Hepatocellular carcinoma or any other malignancy,
4. Hypercoagulable state other than the liver disease related
5. DRUGS- oral contraceptives, anticoagulation or anti-platelet drugs.
6. Child - Pugh C
7. Recent peptic ulcer disease
8. History of Hemorrhagic stroke
9. Pregnancy.
10. Uncontrolled Hypertension
11. Human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Diarrhea | 3 month
  Proportions of patients who will suffer from diarrhea in both groups.
Delayed gastric emptying | 3 month
  Proportions of patients who will suffer from delayed gastric emptying in both groups.

SECONDARY OUTCOMES:
Postoperative complications of the digestive system | 3 month
  Proportions of patients who will suffer from postoperative complications of the digestive system in both groups.
Esophagogastric variceal re-bleeding | 3 month
  Proportions of patients who will suffer from esophagogastric variceal re-bleeding in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dou-Sheng Bai, MD, Study Chair — Clinical Medical College, Yangzhou University; Guo-Qing Jiang, MD, Principal Investigator — Clinical Medical College, Yangzhou University; Ping Chen, MD, Study Director — Clinical Medical College, Yangzhou University
Locations (1):
- Clinical Medical College, Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bai DS, Jin SJ, Zhou BH, Xiang XX, Qian JJ, Zhang C, Gao TM, Jiang GQ. Vagus nerve-guided (modified Bai-Jiang-style) robotic-assisted laparoscopic splenectomy and azygoportal disconnection. Int J Med Robot. 2023 Apr;19(2):e2490. doi: 10.1002/rcs.2490. Epub 2022 Dec 11. PMID 36478144